CLINICAL TRIAL: NCT01883219
Title: Tyrosine Kinase Inhibitor Therapy Based on Molecular Monitoring of BCR/ABL Transcript Levels in Allogeneic Hematopoietic Stem Cell Transplant Recipients With Philadelphia Chromosome-positive Acute Lymphoblastic Leukemia
Brief Title: TKI Therapy Based on Molecular Monitoring in Allogeneic-HSCT Recipients With Philadelphia Chromosome-positive Acute Lymphoblastic Leukemia
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Nanfang Hospital, Southern Medical University (Other)
Collaborators: Peking University People's Hospital (Other); Guangxi Medical University (Other); Guangdong Provincial People's Hospital (Other); Guangzhou General Hospital of Guangzhou Military Command (Other); Sun Yat-Sen Memorial Hospital of Sun Yat-Sen University (Other); Third Affiliated Hospital, Sun Yat-Sen University (Other)
Responsible Party: Principal Investigator, Qifa Liu, Professor, Nanfang Hospital, Southern Medical University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NFEC-201304-K2
Record Dates: First submitted 2013-06-14; First posted 2013-06-21 (Estimated); Last update posted 2017-11-08 (Actual); Status verified 2013-06

CONDITIONS: Philadelphia Chromosome Positive Acute Lymphocytic Leukemia; Stem Cell Transplantation; Minimal Residual Disease
Keywords: Philadelphia chromosome; Acute lymphoblastic leukemia; Allogeneic hematopoietic cell transplantation; Minimal residual disease; Tyrosine kinase inhibitor
MeSH Terms: conditions — Neoplasm, Residual; Philadelphia Chromosome; Precursor Cell Lymphoblastic Leukemia-Lymphoma

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- TKI therapy (Experimental): Treatment with TKI will be initiated if the level of BCR-ABL transcript in the bone marrow is detectable and transcript levels increased for two consecutive tests. TKIs will be given for patients without BCR/ABL mutations and sensitive TKIs will be given for those with mutations.
  Interventions: Drug: TKIs

INTERVENTIONS:
Drug: TKIs — Imatinib was given at a dose of 400mg/d or 600mg/d, dasatinib at a dose of 100mg/d or 140mg/d, and nilotinib at a dose of 400mg twice daily. If the patients had T315I mutations, ponatinib will be given. If the BCR/ABL levels increased or did not decrease after one month's use of TKI, donor lymphocyte infusion will be given and the TKI drugs will be modulated. If the patients experienced hematologic relapse, they will withdraw from the study.

SUMMARY:
The purpose of this study is to evaluate the efficacy of tyrosine kinase inhibitor(TKI) therapy based on molecular monitoring of BCR/ABL levels in Philadelphia chromosome-positive acute lymphoblastic leukemia (Ph+ ALL)undergoing allogeneic hematopoietic stem cell transplantation(allo-HSCT).

DETAILED DESCRIPTION:
Philadelphia chromosome (Ph) is a reciprocal chromosomal translocation t(9;22）(q34;q11), which leads to the formation of the BCR/ABL oncogene. Ph is the most frequent cytogenetic abnormality in ALL characterized by poor outcome. With the BCR/ABL protein TKI, imatinib, in the combination chemotherapy regimes for newly diagnosed Ph+ ALL, more than 95% of patients can achieve complete remission(CR). Several studies have shown decreased relapse rates and improved disease-free survival for patients with imatinib-based treatment prior to allo-HSCT. However, the efficacy of maintenance therapy with imatinib after transplant for Ph+ ALL patients is still uncertain. In addition, acquired resistance to imatinib is frequently caused by point mutations in BCR/ABL that inactivate imatinib.

Detection of minimal residual disease (MRD) after transplant is associated with an increased risk of relapse. Reverse transcription-polymerase chain reaction (RT-PCR) is a sensitive method for detecting low-level BCR/ABL transcripts to assess MRD in Ph+ ALL. It has been corroborated by several reports that detection of MRD after SCT was predictive of imminent relapse.

In this study, we will evaluate the safety and efficacy of TKI therapy, when initiating treatment based on BCR-ABL transcript levels after allo-HSCT.

ELIGIBILITY:
Inclusion Criteria:

* A patient age of 14-65 years
* Allo-HSCT recipient with ph+ ALL
* Subjects (or their legally acceptable representatives) must have signed an informed consent document indicating that they understand the purpose of and procedures required for the study and are willing to participate in the study.

Exclusion Criteria:

* Any abnormality in a vital sign (e.g., heart rate, respiratory rate, or blood pressure)
* patients with hematological relapse, extramedullary involvement of leukemia
* Patients with any conditions not suitable for the trial (investigators' decision)

Ages: 14 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2013-06; Primary Completion 2016-06 (Actual); Study Completion 2017-11 (Estimated)

PRIMARY OUTCOMES:
Overall survival(OS) | 2 years
  OS is defined as continuous survival until death from any cause after HSCT.

SECONDARY OUTCOMES:
Relapse rate | 2 years
  A post-transplant relapse is defined as hematological relapse, extramedullary involvement of leukemia and cytogenetic relapse.
Disease-free survival(DFS) | 2 years
  DFS is defined as continuous survival without relapse or death from any cause after HSCT.
Safety of TKI therapy | 2 years
  The toxicity of TKI is assessed according to the Common Toxicity Criteria, version 3.0.

CONTACTS AND LOCATIONS:
Overall Officials: Qifa Liu, MD, Principal Investigator — Nanfang Hospital, Southern Medical University
Locations (1):
- Department of Hematology,Nanfang Hospital, Southern Medical University, Guangzhou, Guangdong, China

REFERENCES:
- [Background] Yanada M, Sugiura I, Takeuchi J, Akiyama H, Maruta A, Ueda Y, Usui N, Yagasaki F, Yujiri T, Takeuchi M, Nishii K, Kimura Y, Miyawaki S, Narimatsu H, Miyazaki Y, Ohtake S, Jinnai I, Matsuo K, Naoe T, Ohno R; Japan Adult Leukemia Study Group. Prospective monitoring of BCR-ABL1 transcript levels in patients with Philadelphia chromosome-positive acute lymphoblastic leukaemia undergoing imatinib-combined chemotherapy. Br J Haematol. 2008 Nov;143(4):503-10. doi: 10.1111/j.1365-2141.2008.07377.x. PMID 18986386
- [Background] Wassmann B, Pfeifer H, Stadler M, Bornhauser M, Bug G, Scheuring UJ, Bruck P, Stelljes M, Schwerdtfeger R, Basara N, Perz J, Bunjes D, Ledderose G, Mahlberg R, Binckebanck A, Gschaidmeier H, Hoelzer D, Ottmann OG. Early molecular response to posttransplantation imatinib determines outcome in MRD+ Philadelphia-positive acute lymphoblastic leukemia (Ph+ ALL). Blood. 2005 Jul 15;106(2):458-63. doi: 10.1182/blood-2004-05-1746. Epub 2005 Apr 7. PMID 15817679
- [Derived] Liu H, Xuan L, Lin R, Deng L, Fan Z, Nie D, Li X, Liang X, Xu D, Zhang Y, Xu N, Ye J, Jin H, Lin D, Ma L, Sun J, Huang F, Liu Q. A new pre-emptive TKIs strategy for preventing relapse based on BCR/ABL monitoring for Ph+ALL undergoing allo-HCT: a prospective clinical cohort study. Leukemia. 2021 Jul;35(7):2054-2063. doi: 10.1038/s41375-020-01090-4. Epub 2020 Nov 17. PMID 33204013